CLINICAL TRIAL: NCT01199991
Title: Comparison of Xtreme CT and DXA Bone Densitometry
Status: Terminated | Type: Observational
Why Stopped: Limited funding, change in research priorities.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joel S. Finkelstein, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2010P000462
Record Dates: First submitted 2010-09-07; First posted 2010-09-13 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Bone Density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Normative database

SUMMARY:
Dual-energy x-ray absorptiometry (DXA) is currently the most widely used tool for determining bone density. However, most experts consider DXA an imperfect and intermediate technology. DXA is subject to artifact from arthritis and body composition, and also cannot account for geometric or material properties of bone which are also important components of bone strength.

Xtreme CT (high-resolution peripheral quantitative computed tomography, HR-pQCT) is a new technology with dramatically improved spatial resolution. It is able to define bones' cortical and trabecular surfaces in a three-dimensional manner, and therefore provides information on bone microarchitecture as well as bone density. As such, it may provide new information about characteristics of bone strength.

The purpose of this study is to compare Xtreme CT to DXA measurements of bone density, and also to generate a normative database of healthy young adults. This cross-sectional study involves a single visit where both Xtreme CT and DXA measurements will be obtained for a single time-point. This normative database will allow us to generate clinically relevant comparisons between the two imaging technologies.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 20-40 years

Exclusion Criteria:

* Pregnancy
* History of bone modifying diseases (hyperparathyroidism, Paget's, hyperthyroidism, renal failure, nephrolithiasis, liver disease, eating disorder)
* History of amenorrhea
* Use of chronic steroids for >3 months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-08; Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Xtreme CT | single measurement at baseline
  Bone imaging of forearm and lower leg
DXA | single measurement at baseline
  Bone imaging of spine, hip, total body, and forearm

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Finkelstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States